CLINICAL TRIAL: NCT06157489
Title: Effect of Kinesio Tape on Oral and Pharangeal Swallowing Phases in Children With Spastic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Samy Abd Elaziz Alawy, Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 004448
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Dysphagia, Oropharyngeal, Cerebral Palsy
MeSH Terms: conditions — Deglutition Disorders; Cerebral Palsy | interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Active Comparator: Kinesiotape Group In active group, KT was applied in masseter muscle, orbicularis oris and infrahyoid muscles for facilitating suprahyoid muscle and oral sensorimotor exercise In sham group will receive the oral sensorimotor exercise only
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Hamza (Active Comparator)
  Interventions: Other: Kinesio tape
- Noor mohamed (Sham Comparator)
  Interventions: Other: Kinesio tape
- Janna ahmed (Active Comparator)
  Interventions: Other: Kinesio tape
- Hamza salah (Active Comparator)
  Interventions: Other: Kinesio tape
- Mohammed asel (Sham Comparator)
  Interventions: Other: Kinesio tape
- Ali ahmed (Active Comparator)
  Interventions: Other: Kinesio tape
- Malek Mohamed (Sham Comparator)
  Interventions: Other: Kinesio tape
- Sayed Mohamed (Active Comparator)
  Interventions: Other: Kinesio tape
- Omar ahmed (Active Comparator)
  Interventions: Other: Kinesio tape
- Ahmed Mohamed (Sham Comparator)
  Interventions: Other: Kinesio tape
- Yousef salah (Sham Comparator)
  Interventions: Other: Kinesio tape
- Rofan ahmed (Active Comparator)
  Interventions: Other: Kinesio tape
- Kinesio tape hasnot assigned to arm group Exercise only (Sham Comparator)
  Interventions: Other: Kinesio tape
- Fareda salah (Active Comparator)
  Interventions: Other: Kinesio tape
- Abd elrahman ahmed (Active Comparator)
  Interventions: Other: Kinesio tape

INTERVENTIONS:
Other: Kinesio tape — Kinesiotape is applied on masseter muscle, orbi and infrahyoid muscles for facilitating suprahyoid muscle

SUMMARY:
The purpose of current study is to investigate the effect of kinesio tape in children with spastic cerebral palsy having oropharyngeal dysphagia

DETAILED DESCRIPTION:
The study tageted rhe children with spastic cerebral palsy from both sexes will be selected from hospital of Tanta university

Inclusion criteria:

1. Age ranges from 2 to 7 years.
2. The degree of dysphagia ranges from 4 to 6 level according to functional oral intake scale (appendix II).
3. Diagnosed as spastic diplegia or quadriplegia.
4. Able to understand and follow instructions.

Exclusion criteria:

Children will be excluded if they have any of the following criteria:

1. Severe visual and auditory problems.
2. History of maxillary, head or neck surgical procedures.
3. Botulinum toxin treatment of upper esophageal sphincter dysfunction, esophageal dysphagia and/or gastroesophageal reflux disease during the previous six months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranges from 3 to 7 years.
2. The degree of dysphagia ranges from 4 to 6 level according to functional oral intake scale (appendix II).
3. Diagnosed as spastic diplegia or quadriplegia.
4. Able to understand and follow instructions.

Exclusion Criteria:

Children will be excluded if they have any of the following criteria:

1. Severe visual and auditory problems.
2. History of maxillary, head or neck surgical procedures.
3. Botulinum toxin treatment of upper esophageal sphincter dysfunction, esophageal dysphagia and/or gastroesophageal reflux disease during the previous six months.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Oral motor assessment sacle | 1 month
  Assessment for oral phase

SECONDARY OUTCOMES:
ultrasonography | 1 month
  Assessment of pharangal phase

CONTACTS AND LOCATIONS:
Locations (1):
- Hadeer samy abd elaziz, Tanta, Egypt